CLINICAL TRIAL: NCT03450473
Title: A Prospective Case Series Evaluating Surgimend Mp® In Patients Undergoing Complex Abdominal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WU001 Surgimend Mp®
Record Dates: First submitted 2018-01-08; First posted 2018-03-01 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-01

CONDITIONS: Hernia, Ventral
Keywords: Mesh
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SurgiMend® MP (Other): Patients will not be randomized as this is a case series study involving the evaluation of only 1 type of mesh (SurgiMend MP®).
  Interventions: Device: SurgiMend® MP

INTERVENTIONS:
Device: SurgiMend® MP — SurgiMend MP® is an acellular dermal tissue matrix derived from bovine dermis. The device is supplied sterile in a variety of sizes to be trimmed by the surgeon to meet the individual patient's needs. SurgiMend MP® will be used for abdominal wall reinforcement in patients with complex ventral hernia repair.

SUMMARY:
Large abdominal wall hernias are surgically challenging to repair and often associated with significant postoperative complications. Risk factors associated with surgical site complications, such as infection and wound dehiscence, include obesity, diabetes, and smoking. In these high risk patients, the placement of synthetic mesh increases the risk of mesh infection, enterocutaneous fistula formation, and mesh explantation. One of the larger studies of risk factors associated with mesh explantation demonstrated concomitant intra-abdominal procedures have a greater than 6-fold increased hazard of subsequent mesh explantation. As an alternative to synthetic meshes, bioprosthetic meshes derived from the decellularization and processing of allogeneic or xenogeneic tissue sources have been introduced that can often allow the surgeon to treat the surgical site occurrences and salvage the repair without required mesh explantation. Low rates of mesh infection and explantation have been reported for bioprosthetic meshes and are recommended in these complicated patients by the Ventral Hernia Working Group, based on the best available clinical evidence. Despite widespread use of bioprosthetic mesh, there continues to be concern for complications associated with their use (i.e. high seroma and recurrence rates, etc.). This has led to the modification of these matrices by several industry leaders (Acelity, Cook, Integra, etc.) to include a fenestrated platform to allow for fluid to flow through the matrix upon implantation while supporting regeneration in complex abdominal wall reconstruction. To our knowledge, there are no clinical studies prospectively evaluating the long term clinical outcomes for abdominal wall reconstruction procedures involving fenestrated macropourous biologic matrices.This macroporous technology allows for tissue revascularization and integration of the biologic graft and thus an expected improvement in overall outcome. Bioprosthetic fenestrated materials such as Surgimend MP® were developed to assist with earlier incorporation and vascularization of the biologic graft while providing reinforcement of hernia repair. However, there is an absence of high quality prospective data regarding the use of these materials in complicated abdominal wall reconstruction, and no comparative data exists.

This study is a prospective, case series study evaluating the efficacy and performance of SurgiMend MP® during complex ventral hernia repairs. This case series involves a biologically derived hernia mesh under its cleared FDA indication for hernia repair. Efficacy will be determined by quantifying surgical complications, hernia recurrence, and cost effectiveness endpoints.

DETAILED DESCRIPTION:
Large abdominal wall hernias are surgically challenging to repair and often associated with significant postoperative complications. Risk factors associated with surgical site complications, such as infection and wound dehiscence, include obesity, diabetes, and smoking. In these high risk patients, the placement of synthetic mesh increases the risk of mesh infection, enterocutaneous fistula formation, and mesh explantation. One of the larger studies of risk factors associated with mesh explantation demonstrated concomitant intra-abdominal procedures have a greater than 6-fold increased hazard of subsequent mesh explantation. As an alternative to synthetic meshes, bioprosthetic meshes derived from the decellularization and processing of allogeneic or xenogeneic tissue sources have been introduced that can often allow the surgeon to treat the surgical site occurrences and salvage the repair without required mesh explantation. Low rates of mesh infection and explantation have been reported for bioprosthetic meshes and are recommended in these complicated patients by the Ventral Hernia Working Group, based on the best available clinical evidence. Despite widespread use of bioprosthetic mesh, there continues to be concern for complications associated with their use (i.e. high seroma and recurrence rates, etc.). This has led to the modification of these matrices by several industry leaders (Acelity, Cook, Integra, etc.) to include a fenestrated platform to allow for fluid to flow through the matrix upon implantation while supporting regeneration in complex abdominal wall reconstruction. To our knowledge, there are no clinical studies prospectively evaluating the long term clinical outcomes for abdominal wall reconstruction procedures involving fenestrated macropourous biologic matrices.This macroporous technology allows for tissue revascularization and integration of the biologic graft and thus an expected improvement in overall outcome. Bioprosthetic fenestrated materials such as Surgimend MP® were developed to assist with earlier incorporation and vascularization of the biologic graft while providing reinforcement of hernia repair. However, there is an absence of high quality prospective data regarding the use of these materials in complicated abdominal wall reconstruction, and no comparative data exists.

This study is a prospective, case series study evaluating the efficacy and performance of SurgiMend MP® during complex ventral hernia repairs. This case series involves a biologically derived hernia mesh under its cleared FDA indication for hernia repair. Efficacy will be determined by quantifying surgical complications, hernia recurrence, and cost effectiveness endpoints.

Subjects will be identified by the investigators and/or personnel assigned by the investigators, as patients with large complex ventral hernia expected to be repaired with bioprosthetic mesh.

Subjects will have a baseline visit where they will have a physical exam and complete quality of life questionnaires and a pain scale. Photographs will be taken at this visit as well. Demographic and medical and surgical history will be collected. The investigators will then assess the subject intra-operatively to confirm the need and appropriate placement of SurgiMend mesh. The subjects that have mesh placed will be followed at hospital discharge, 3 months, 6 months, and 12 months to assess for changes in health, adverse events, questionnaire completion, and evaluation of surgical site for complications and recurrence. The visits may take place by phone if the subject cannot return to clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥ 18 years of age and able to give their own consent.
2. The subject is able and willing to comply with study procedures and a signed and dated informed consent is obtained.
3. The subject has a complex ventral hernia
4. The surgeon intends to use bioprosthetic mesh in the repair of the hernia
5. The hernia meets the definition of complex.

   For this study a hernia defect will be considered complex if:

   5.1. a hernia defect is large enough to require component separation to achieve midline fascial closure under physiologic tension 5.2. or the surgical wound is class II -potentially contaminated or class III - contaminated without signs of infection as defined by the CDC wound classification (see Table 1) 5.3. or a patient classified as at risk for surgical site complications by having 2 or more of the following comorbidities:
   * Current smoker or recent history of smoking
   * Obesity (BMI ≥ 30)
   * Type I or Type II diabetes
   * Chronic Obstructive Pulmonary Disease (COPD)
   * Poor nutritional status as judged by the Investigator
   * Current immunosuppressive therapy
   * Current and/or recent (within 30 days of planned surgery) Corticosteriod use
   * Prior Mesh infection
6. Life expectancy of the patient is considered by the physician to be greater than at least 1 year
7. The subject has no known hypersensitivity to bovine collagen
8. The subject has no obvious condition interfering with their ability to comply with the treatment regimen
9. The subject is willing and capable of returning for all follow-up evaluations, in the opinion of the treating physician

Exclusion Criteria:

Pre-Operative Exclusion:

1. < 18 years of age
2. Have abdominal loss of domain such that the operation would be impractical or would adversely affect respiratory or cardiovascular function to an unacceptable degree in the opinion of the Investigator
3. Participation in an investigational drug or device study within the past 6 weeks prior to enrollment into this trial
4. Have a known collagen metabolism disorder or any medical condition that could interfere with normal tissue healing process as determined by the Investigator

Intra-Operative Exclusion Criteria:

Subjects will be excluded from the study after the index operation if any of the following exclusion criteria are met:

1. Primary closure of the skin and subcutaneous tissue is not achieved at the index operation
2. Bioprosthetic mesh was not used in the repair for any reason
3. Primary Fascial closure unable to be obtained i.e. bridged closure
4. Unable to place the mesh in the retrorectus space (no intraperitoneal placement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant Bochicchio, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SurgiMend® MP
Started | 24
Completed | 20
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | SurgiMend® MP
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15
  African American | 5

OUTCOME MEASURES:

1. Primary Outcome: The Frequency of Hernia Recurrence Diagnosed by Physical Exam or CT Scan (if Clinically Indicated)
Description: The frequency of hernia recurrence diagnosed by physical exam or CT Scan (if clinically indicated)
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | SurgiMend® MP
Number analyzed (Participants) | 20
Participants | 1

ADVERSE EVENTS:
Time Frame: For the purpose of this post-market case series study, only adverse events or serious adverse events that were related to the surgical procedure or device were recorded. The collection of AE's began immediately after the patient had mesh surgically implanted. AEs that occurred from surgery through completion of the final follow-up visit (36 months) were collected.
Description: For the purpose of this post-market case series study, only adverse events or serious adverse events that were related to the surgical procedure or device were recorded.
Arm/Group | SurgiMend® MP
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 6/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SurgiMend® MP (N=20)
Seroma (Surgical and medical procedures) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SurgiMend® MP (N=20)
Post Operative Pain (Surgical and medical procedures) | 1
Hematoma (Surgical and medical procedures) | 1
Wound Necrosis (Surgical and medical procedures) | 1
Hernia Recurrence (Surgical and medical procedures) | 1
Seroma (Surgical and medical procedures) | 1
Wound Dehiscence (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT03450473/Prot_000.pdf